CLINICAL TRIAL: NCT01106625
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Arm, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin and Sulphonylurea Therapy
Brief Title: The CANTATA-MSU Trial (CANagliflozin Treatment And Trial Analysis - Metformin and SUlphonylurea)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017005; 28431754DIA3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-04-01; First posted 2010-04-20 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Placebo; Metformin; Sulphonylurea; Hemoglobin A1c; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
  Interventions: Drug: Canagliflozin; Drug: Metformin; Drug: Sulphonylruea
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
  Interventions: Drug: Canagliflozin; Drug: Metformin; Drug: Sulphonylruea
- Placebo (Placebo Comparator): Each patient will receive matching placebo once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
  Interventions: Drug: Placebo; Drug: Metformin; Drug: Sulphonylruea

INTERVENTIONS:
Drug: Canagliflozin — One 100 mg or 300 mg over-encapsulated tablet orally (by mouth) once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg
Drug: Placebo — One matching placebo capsule orally once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
  Arms: Placebo
Drug: Metformin — The patient's stable dose of background metformin therapy should be continued throughout the study.
Drug: Sulphonylruea — The patient's stable dose of background sulphonylurea therapy should be continued throughout the study.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 different doses of canagliflozin compared with placebo in patients with type 2 diabetes mellitus who are receiving treatment with metformin and sulphonylurea and have inadequate glycemic (blood sugar) control.

DETAILED DESCRIPTION:
Canagliflozin is a drug that is being tested to see if it may be useful in treating patients diagnosed with type 2 diabetes mellitus (T2DM). This is a randomized (study drug assigned by chance), double-blind (neither the patient or the study doctor will know the name of the assigned treatment), placebo-controlled, parallel-group, 3-arm (3 treatment groups) multicenter study to determine the efficacy, safety, and tolerability of canagliflozin (100 mg and 300 mg) compared to placebo (a capsule that looks like all the other treatments but has no real medicine) in patients with T2DM who are not achieving an adequate response from current antihyperglycemic therapy with metformin and sulphonylurea to control their diabetes. Approximately 450 patients with T2DM who are receiving treatment with metformin and sulphonylurea and have inadequate glycemic (blood sugar) control will receive once daily treatment with canagliflozin (100 mg or 300 mg) or placebo capsules for 52 weeks (includes 26 weeks of double-blind treatment followed by a 26-week extension period). In addition, all patients will take protocol-specified stable doses of metformin and sulphonylurea for the duration of the study. Patients will participate in the study for approximately 59 to 72 weeks. During the study, if a patient's fasting blood sugar remains high despite treatment with study drug, the patient will receive treatment with insulin (rescue therapy) consistent with local prescribing information. During treatment, patients will be monitored for safety by review of adverse events, results from laboratory tests, 12-lead electrocardiograms (ECGs), vital signs measurements, body weight, physical examinations, and self-monitored blood glucose (SMGB) measurements. The primary outcome measure in the study is to assess the effect of canagliflozin relative to placebo on hemoglobin A1c (HbA1c) after 26 weeks of treatment. Study drug will be taken orally (by mouth) once daily before the first meal each day unless otherwise specified. All patients will take single-blind placebo capsules for 2 weeks before randomization. After randomization, patients will take double-blind canagliflozin (100 mg or 300 mg) or matching placebo for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM and be currently treated with metformin and sulphonylurea
* Patients in the study must have a HbA1c between >=7 and <=10.5%
* Patients must have a fasting plasma glucose (FPG) <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy, or a severe hypoglycemic episode within 6 months before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (76):
- United States (37):
  - Huntsville, Alabama
  - Little Rock, Alaska
  - Phoenix, Arizona
  - Chino, California
  - Fair Oaks, California
  - Roseville, California
  - Wes Hills, California
  - Waterbury, Connecticut
  - Jacksonville, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Roswell, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Reisterstown, Maryland
  - Olive Branch, Mississippi
  - St Louis, Missouri
  - Westfield, New York
  - Greenville, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Altoona, Pennsylvania
  - Harleysville, Pennsylvania
  - Levittown, Pennsylvania
  - Sellersville, Pennsylvania
  - Greer, South Carolina
  - Bryan, Texas
  - Dallas, Texas
  - DeSoto, Texas
  - Salt Lake City, Utah
  - South Burlington, Vermont
  - Wenatchee, Washington
- Australia (5):
  - Freemantle
  - Heidelberg Heights
  - Meadowbrook
  - Nedlands
  - Wollongong
- Belgium (4):
  - Aalst
  - Bonheiden
  - Edegem
  - Leuven
- France (5):
  - Corbeil-Essonnes
  - La Rochelle
  - Le Creusot
  - Poitiers
  - Vénissieux
- Guatemala City, Guatemala
- Hungary (4):
  - Balatonfüred
  - Budapest
  - Győr
  - Zalaegerszeg
- Israel (4):
  - Haifa
  - Holon
  - Jerusalem
  - Tel Aviv
- Mexico (2):
  - Guadalajara
  - Monterrey
- Puerto Rico (2):
  - Carolina
  - Trujillo Alto
- Russia (3):
  - Arkhangelsk
  - Saint Petersburg
  - Samara
- Spain (5):
  - Alicante
  - Almería
  - Málaga
  - Seville
  - Valencia
- United Kingdom (4):
  - Belfast
  - Bolton
  - Liverpool
  - Manchester

REFERENCES:
- [Derived] Cai J, Delahanty LM, Akapame S, Slee A, Traina S. Impact of Canagliflozin Treatment on Health-Related Quality of Life among People with Type 2 Diabetes Mellitus: A Pooled Analysis of Patient-Reported Outcomes from Randomized Controlled Trials. Patient. 2018 Jun;11(3):341-352. doi: 10.1007/s40271-017-0290-4. PMID 29313267
- [Derived] Davies MJ, Merton K, Vijapurkar U, Yee J, Qiu R. Efficacy and safety of canagliflozin in patients with type 2 diabetes based on history of cardiovascular disease or cardiovascular risk factors: a post hoc analysis of pooled data. Cardiovasc Diabetol. 2017 Mar 21;16(1):40. doi: 10.1186/s12933-017-0517-7. PMID 28327140
- [Derived] Pfeifer M, Townsend RR, Davies MJ, Vijapurkar U, Ren J. Effects of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on blood pressure and markers of arterial stiffness in patients with type 2 diabetes mellitus: a post hoc analysis. Cardiovasc Diabetol. 2017 Feb 27;16(1):29. doi: 10.1186/s12933-017-0511-0. PMID 28241822
- [Derived] Gilbert RE, Mende C, Vijapurkar U, Sha S, Davies MJ, Desai M. Effects of Canagliflozin on Serum Magnesium in Patients With Type 2 Diabetes Mellitus: A Post Hoc Analysis of Randomized Controlled Trials. Diabetes Ther. 2017 Apr;8(2):451-458. doi: 10.1007/s13300-017-0232-0. Epub 2017 Feb 14. PMID 28197834
- [Derived] Qiu R, Balis D, Xie J, Davies MJ, Desai M, Meininger G. Longer-term safety and tolerability of canagliflozin in patients with type 2 diabetes: a pooled analysis. Curr Med Res Opin. 2017 Mar;33(3):553-562. doi: 10.1080/03007995.2016.1271780. Epub 2017 Jan 4. PMID 27977934
- [Derived] John M, Cerdas S, Violante R, Deerochanawong C, Hassanein M, Slee A, Canovatchel W, Hamilton G. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus living in hot climates. Int J Clin Pract. 2016 Sep;70(9):775-85. doi: 10.1111/ijcp.12868. PMID 27600862
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Lavalle-Gonzalez FJ, Eliaschewitz FG, Cerdas S, Chacon Mdel P, Tong C, Alba M. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus from Latin America. Curr Med Res Opin. 2016;32(3):427-39. doi: 10.1185/03007995.2015.1121865. Epub 2016 Jan 14. PMID 26579834
- [Derived] Blonde L, Woo V, Mathieu C, Yee J, Vijapurkar U, Canovatchel W, Meininger G. Achievement of treatment goals with canagliflozin in patients with type 2 diabetes mellitus: a pooled analysis of randomized controlled trials. Curr Med Res Opin. 2015 Nov;31(11):1993-2000. doi: 10.1185/03007995.2015.1082991. Epub 2015 Sep 28. PMID 26373629
- [Derived] Gavin JR 3rd, Davies MJ, Davies M, Vijapurkar U, Alba M, Meininger G. The efficacy and safety of canagliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2015;31(9):1693-702. doi: 10.1185/03007995.2015.1067192. Epub 2015 Sep 4. PMID 26121561
- [Derived] Cefalu WT, Stenlof K, Leiter LA, Wilding JP, Blonde L, Polidori D, Xie J, Sullivan D, Usiskin K, Canovatchel W, Meininger G. Effects of canagliflozin on body weight and relationship to HbA1c and blood pressure changes in patients with type 2 diabetes. Diabetologia. 2015 Jun;58(6):1183-7. doi: 10.1007/s00125-015-3547-2. Epub 2015 Mar 27. PMID 25813214
- [Derived] Weir MR, Januszewicz A, Gilbert RE, Vijapurkar U, Kline I, Fung A, Meininger G. Effect of canagliflozin on blood pressure and adverse events related to osmotic diuresis and reduced intravascular volume in patients with type 2 diabetes mellitus. J Clin Hypertens (Greenwich). 2014 Dec;16(12):875-82. doi: 10.1111/jch.12425. Epub 2014 Oct 20. PMID 25329038
- [Derived] Usiskin K, Kline I, Fung A, Mayer C, Meininger G. Safety and tolerability of canagliflozin in patients with type 2 diabetes mellitus: pooled analysis of phase 3 study results. Postgrad Med. 2014 May;126(3):16-34. doi: 10.3810/pgm.2014.05.2753. PMID 24918789
- [Derived] Weir MR, Kline I, Xie J, Edwards R, Usiskin K. Effect of canagliflozin on serum electrolytes in patients with type 2 diabetes in relation to estimated glomerular filtration rate (eGFR). Curr Med Res Opin. 2014 Sep;30(9):1759-68. doi: 10.1185/03007995.2014.919907. Epub 2014 May 22. PMID 24786834
- [Derived] Sinclair A, Bode B, Harris S, Vijapurkar U, Mayer C, Fung A, Shaw W, Usiskin K, Desai M, Meininger G. Efficacy and safety of canagliflozin compared with placebo in older patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. BMC Endocr Disord. 2014 Apr 18;14:37. doi: 10.1186/1472-6823-14-37. PMID 24742013
- [Derived] Polidori D, Mari A, Ferrannini E. Canagliflozin, a sodium glucose co-transporter 2 inhibitor, improves model-based indices of beta cell function in patients with type 2 diabetes. Diabetologia. 2014 May;57(5):891-901. doi: 10.1007/s00125-014-3196-x. Epub 2014 Mar 1. PMID 24585202
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus with inadequate control despite treatment with metformin and sulphonylurea therapy. The study was conducted between 07 April 2010 and 17 April 2012 and recruited patients from 85 study centers in 11 countries worldwide.
Pre-assignment Details: A total of 469 patients were randomly allocated to the 3 treatment arms in the study. All 469 patients received at least 1 dose of study drug and were included in the modified intent-to-treat analysis set (used for the week 26 efficacy analyses). All 469 patients were included in the week 26 and week 52 safety analysis sets.
Groups:
- Placebo: Each patient received matching placebo once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
Period: Core Period: Baseline to Week 26
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 156 | 157 | 156
Completed | 123 | 129 | 129
Not Completed | 33 | 28 | 27
Not completed — Adverse Event | 6 | 8 | 8
Not completed — Lost to Follow-up | 5 | 0 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 3
Not completed — Withdrawal by Subject | 6 | 9 | 7
Not completed — Unable to take rescue therapy | 4 | 1 | 0
Not completed — Creatinine, or eGFR withdrawal criteria | 0 | 1 | 1
Not completed — Noncompliance with study drug | 1 | 1 | 0
Not completed — Other | 8 | 7 | 4
Period: Extension Period: Week 26 to Week 52
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 119 (4 pts discontinued last day of core: physician decision (1), noncompliance (1), not specified (2).) | 127 (2 pts discontinued last day of core: adverse event (1), not specified (1).) | 128 (1 pt discontinued last day of core: withdrawal by subject (1).)
Completed | 90 | 109 | 111
Not Completed | 29 | 18 | 17
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Unable to take rescue therapy | 14 | 5 | 4
Not completed — Creatinine or eGFR withdrawal criteria | 1 | 1 | 2
Not completed — Other | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 156 | 157 | 156 | 469
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 130 | 121 | 134 | 385
  >=65 years | 26 | 36 | 22 | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 56.7 (8.36) | 57.3 (10.47) | 56 (8.95) | 56.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 81 | 69 | 230
  Male | 76 | 76 | 87 | 239
Region of Enrollment [Number; unit: participants]
  AUSTRALIA | 3 | 6 | 4 | 13
  BELGIUM | 3 | 1 | 6 | 10
  FRANCE | 4 | 7 | 9 | 20
  GUATEMALA | 15 | 12 | 16 | 43
  HUNGARY | 11 | 14 | 11 | 36
  ISRAEL | 1 | 6 | 8 | 15
  MEXICO | 11 | 11 | 11 | 33
  RUSSIAN FEDERATION | 14 | 13 | 8 | 35
  SPAIN | 5 | 7 | 8 | 20
  UNITED KINGDOM | 8 | 6 | 5 | 19
  UNITED STATES | 81 | 74 | 70 | 225

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 26 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin once daily for for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 150 | 155 | 152
Percent | -0.13 (0.075) | -0.85 (0.075) | -1.06 (0.076)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.71, 95% CI 2-sided [-0.904 to -0.524], Standard Error of Mean 0.097
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.92, 95% CI 2-sided [-1.114 to -0.732], Standard Error of Mean 0.097

2. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 26
Description: The table below shows the percentage of patients with HbA1c<7% at Week 26 in each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 150 | 155 | 152
Percentage of patients | 18 | 43.2 | 56.6
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.42, 95% CI 2-sided [2.48 to 7.87]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.80, 95% CI 2-sided [4.86 to 15.95]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 150 | 155 | 152
mg/dL | 4.11 (3.629) | -18.2 (3.629) | -30.5 (3.650)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -22.3, 95% CI 2-sided [-31.53 to -13.16], Standard Error of Mean 4.627
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -34.6, 95% CI 2-sided [-43.86 to -25.42], Standard Error of Mean 4.692

4. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 150 | 156 | 154
Percent change | -0.7 (0.3) | -2.1 (0.3) | -2.6 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.4, 95% CI 2-sided [-2.1 to -0.7], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.0, 95% CI 2-sided [-2.7 to -1.3], Standard Error of Mean 0.4

5. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 150 | 156 | 154
mmHg | -2.65 (0.982) | -4.89 (0.976) | -4.27 (0.980)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.077, ANCOVA; Least-Squares Mean Difference = -2.24, 95% CI 2-sided [-4.719 to 0.241], Standard Error of Mean 1.262
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.201, ANCOVA; Least-Squares Mean Difference = -1.62, 95% CI 2-sided [-4.111 to 0.866], Standard Error of Mean 1.266

6. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in triglycerides from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 134 | 145 | 142
Percent change | 11.6 (4.2) | 5.4 (4.2) | 8.5 (4.2)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.256, ANCOVA; Least-Squares Mean Difference = -6.2, 95% CI 2-sided [-16.9 to 4.5], Standard Error of Mean 5.4
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.571, ANCOVA; Least-Squares Mean Difference = -3.1, 95% CI 2-sided [-13.8 to 7.6], Standard Error of Mean 5.5

7. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in HDL-C from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 135 | 145 | 141
Percent change | 3.2 (1.3) | 5.7 (1.3) | 6.5 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.153, ANCOVA; Least-Squares Mean Difference = 2.5, 95% CI 2-sided [-0.9 to 5.9], Standard Error of Mean 1.7
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.056, ANCOVA; Least-Squares Mean Difference = 3.4, 95% CI 2-sided [-0.1 to 6.8], Standard Error of Mean 1.8

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 52 weeks.
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Groups:
- Placebo: Baseline to Week 26: Each patient received matching placebo once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea. Data are presented for Baseline to Week 26.
- Canagliflozin 100 mg: Baseline to Week 26: Each patient received 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea. Data are presented for Baseline to Week 26.
- Canagliflozin 300 mg: Baseline to Week 26: Each patient received 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea. Data are presented for Baseline to Week 26.
- Placebo: Baseline to Week 52: Each patient received matching placebo once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea. Data are presented for Baseline to Week 52.
- Canagliflozin 100 mg: Baseline to Week 52: Each patient received 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea. Data are presented for Baseline to Week 52.
- Canagliflozin 300 mg: Baseline to Week 52: Each patient received 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea. Data are presented for Baseline to Week 52.
Arm/Group | Placebo: Baseline to Week 26 | Canagliflozin 100 mg: Baseline to Week 26 | Canagliflozin 300 mg: Baseline to Week 26 | Placebo: Baseline to Week 52 | Canagliflozin 100 mg: Baseline to Week 52 | Canagliflozin 300 mg: Baseline to Week 52
Serious Adverse Events (participants affected / at risk) | 9/156 | 5/157 | 6/156 | 13/156 | 7/157 | 8/156
Other Adverse Events (participants affected / at risk) | 31/156 | 42/157 | 38/156 | 52/156 | 63/157 | 54/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Baseline to Week 26 (N=156) | Canagliflozin 100 mg: Baseline to Week 26 (N=157) | Canagliflozin 300 mg: Baseline to Week 26 (N=156) | Placebo: Baseline to Week 52 (N=156) | Canagliflozin 100 mg: Baseline to Week 52 (N=157) | Canagliflozin 300 mg: Baseline to Week 52 (N=156)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Uterine enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 0 | 1 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Ulcer haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Gangrene (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Lobar pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Scrotal gangrene (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Baseline to Week 26 (N=156) | Canagliflozin 100 mg: Baseline to Week 26 (N=157) | Canagliflozin 300 mg: Baseline to Week 26 (N=156) | Placebo: Baseline to Week 52 (N=156) | Canagliflozin 100 mg: Baseline to Week 52 (N=157) | Canagliflozin 300 mg: Baseline to Week 52 (N=156)
Influenza (Infections and infestations) | 0 | 0 | 0 | 8 | 4 | 8 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3 | 8 | 3 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 8 | 8 | 8 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Headache (Nervous system disorders) | 0 | 0 | 0 | 5 | 11 | 2 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 10 | 5 | 8 | 11 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Nasopharyngitis (Infections and infestations) | 4 | 6 | 8 | 10 | 9 | 9 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Upper respiratory tract infection (Infections and infestations) | 10 | 17 | 6 | 13 | 21 | 9 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Urinary tract infection (Infections and infestations) | 8 | 9 | 7 | 12 | 12 | 9 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 8 | 8 | 2 | 9 | 8 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 11 | 9 | 9 | 13 | 11 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.